CLINICAL TRIAL: NCT00973440
Title: Computer-Based Comprehensive Geriatric Assessment in Oncology for Individuals 70 or Older With Colorectal, Breast or Lung Cancer
Brief Title: Computer-Based Comprehensive Geriatric Assessment in Oncology for Individuals 70 or Older With Gastrointestinal Malignancies
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Nadine A. Jackson, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 09-035
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Rectal Cancer; Breast Cancer; Lung Cancer
Keywords: geriatric assessment
MeSH Terms: conditions — Rectal Neoplasms; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Older individuals account for one-third of new cancer cases and cancer-related deaths in the United States. Older individuals are more susceptible to having a decrease in physical and mental function following chemotherapy treatment. Geriatric assessment may provide a way to identify those older individuals at greatest risk of functional decline before treatment starts and during the period of treatment. Geriatric assessment includes a set of screening questions and tests designed to determine the physical and mental status of the individual at a point in time. Geriatric assessment also includes review of medications and other medical conditions the individual may have that may affect function. The investigators are conducting this study to determine if older individuals are able to complete the geriatric assessment using a computer format and how that corresponds to their treating physician's assessment of their functional status before and after starting a new chemotherapy treatment for colon, rectal, breast or lung cancer. The investigators will also evaluate the usefulness of a computerized form of geriatric assessment.

DETAILED DESCRIPTION:
* Participants will complete the geriatric assessment on the computer either at their home via the web (if they have internet access) or in the clinic at their next visit prior to seeing the doctor.
* All individuals will have a unique way to sign on to the computer program that protects the information so that only the participant and the research team will be able to view it. Individuals who require assistance to answer the questions will have help provided by a research assistant.
* We will ask participants to complete the geriatric assessment a second time at 4 months after they have enrolled on the study or 1 month after completing their chemotherapy treatment, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients with colorectal, breast or lung cancer at any stage who are under consideration for initiation of or change in cytotoxic chemotherapy regimen. Patients must start chemotherapy within 4 weeks of enrollment. Chemotherapy regimens may include traditional cytotoxic therapy, oral biological agent, or combination of a biologic therapy and cytotoxic chemotherapy.
* Patients age 70 or older at enrollment
* Patients must be able to read English and able to complete the web-based computer questionnaire

Exclusion Criteria:

* Patients with a physical limitation preventing computer use (visual impairment, inability to use computer mouse or touch screen).
* Patients who are hospitalized or enrolled in hospice

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants are identified by review of the clinic visit schedule at the Dana-Farber Cancer Institute, identifying individuals age 70 and older diagnosed with colon, rectal, breast or lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and added clinical utility of a self-administered computer-based version of an abbreviated comprehensive geriatric assessment tool. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nadine J McCleary, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States